CLINICAL TRIAL: NCT02399891
Title: Acute Myocardial Infarction Quality Assurance Project
Acronym: AMIQA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Derek Exner (Other)
Responsible Party: Sponsor-Investigator, Dr. Derek Exner, Professor, University of Calgary
Organization: University of Calgary (Other)
Other Study IDs: QA20111211
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Myocardial Infarction; Death; Heart Failure
Keywords: Remodeling; Prognosis; Incidence; Quality Assurance; Ejection Fraction; Sudden Death
MeSH Terms: conditions — Myocardial Infarction; Death; Heart Failure; Death, Sudden | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective: MI prior to December 11, 2011
  Interventions: Other: Standard of Care
- Prospective: MI on or after December 11, 2011
  Interventions: Other: Quality Assurance Implementation

INTERVENTIONS:
Other: Quality Assurance Implementation
  Groups: Prospective
Other: Standard of Care
  Groups: Retrospective

SUMMARY:
Cohort study aimed at evaluating the incidence of left ventricular (LV) dysfunction after myocardial infraction (MI) and assessing the prognostic utility of change in ejection fraction (EF) over the initial 12 months after MI.

DETAILED DESCRIPTION:
Background

Patients suffering a myocardial infraction (MI) may have from minimal to extensive myocardial damage. While severe left ventricular (LV) dysfunction that persists beyond the initial 2-3 months of an MI is a predictor of sudden death, the prognostic significance of less severe LV dysfunction after MI is unclear.

There is significant clinical value in quantifying LV function after the recovery phase of an MI. This information is vital in guiding the breadth and duration of therapies known to improve prognosis (beta-blockers, ACE inhibitors, angiotensin blockers, anticoagulants, and others). Further, it will identify patients in whom other therapies, such as an implantable cardioverter defibrillator (ICD), are recommended. Yet, no guidelines to guide clinical decision making in terms of collecting follow-up ejection fraction (EF) data in such patients who do not also have overt heart failure.

Purpose The Acute Myocardial Infarction Quality Assurance (AMIQA) project proposes to

1. document clinical practice by collecting data on the proportion of patients with initial LV dysfunction after MI without a follow-up EF assessment arranged,
2. collect follow-up EF data in patients with initial LV dysfunction post-MI and evaluate the prognostic significant of EF early and late after MI as well as factors associated with the change in value, and
3. educate physicians regarding the importance of EF reassessment after MI.

Follow up LV assessment

The current guidelines do not clearly provide clear indications to the appropriate timing or modality of follow up left ventricular assessments. We have chosen to define an adequate follow up LV assessment to occur within 2 to 12 months post-myocardial infarction, measured by any modality such as echocardiography, cardiac MRI, or nuclear perfusion scan.

Overall Study Objectives

1. To evaluate the relationship of changes in EF after MI with clinical variables such as age, gender, co-morbid conditions, MI characteristics, and the prescription of pharmacological agents after MI.
2. To assess the relationship of changes in EF after MI with clinical outcomes.

Study Methodology and Data Collection

This study will be conducted in three phases:

1. determining the existing practice of assessing left ventricular ejection fraction following myocardial infarction within the Calgary region (Quality Assurance);
2. determining the factors associated with LVEF improvement, stability and decline post-MI and the relationship of these with outcome (Prognostic Factor Study);
3. educating the clinical community about the importance of follow up LVEF assessments and reporting the findings of this through presentations, educational materials and/or academic publications (Knowledge Dissemination)

Study Population

The study population will include patients presenting with an acute myocardial infarction (NSTEMI or STEMI) undergoing cardiac catheterization at the Foothills Medical Center, who have significant left ventricular impairment upon initial LV assessment as defined as at least:

* At least mod dysfunction (LVEF < 0.40) if no prior history of MIs (i.e. first MI)
* More than mild-moderate dysfunction (LVEF < 0.45) if prior history of MI Exclusion criteria include: patients lost to follow up by their family physician or primary cardiologist, and patients who are deceased who do not have a follow-up EF.

Patients will be identified using the APPROACH (Alberta Provincial Project for Outcome Assessment in Coronary Heart Disease (www.approach.org)) database. All patients will have provided written, informed consent as part of their participation in APPROACH.

AMIQA Phase I: Quality Assurance

Part One (Quality Assurance) will include patients with an MI occurring between July 1, 2010 to November 30, 2011 (15 months). The list of patients who have had myocardial infarctions undergoing cardiac catheterization at the Foothills Medical Center between these dates can be obtained through the APPROACH database. For the patients that meet the initial inclusion criteria for significant LV dysfunction post-MI, the study group will determine if a follow up LVEF assessment has been performed within 2 to 12 months post-MI by contacting the patient's family physician and/or primary cardiologist for any records of LVEF measurements, and searching through the following electronic databases.

AMIQA Phase II: Prognostic Factor Study

Part Two (Prognostic Factor Study) will include patients with myocardial infarctions occurring on December 5, 2011 until December 5, 2012 (12 months). The list of patients who have had myocardial infarctions undergoing cardiac catheterization at the Foothills Medical Center between these dates can be obtained through the APPROACH database. For the patients that meet the initial inclusion criteria for significant LV dysfunction post-MI (as described in section 5.1), the study group will contact the patient, the patient's family physician, and/or patient's primary cardiologist to order a follow up LVEF measurement within 2 to 12 months post- myocardial infarction. That is, all patients that have significant LV dysfunction will undergo follow up LVEF measurements between December 5, 2011 and December 5, 2012. Modalities for follow up LVEF measurements will include echocardiogram, cardiac MRI, and nuclear perfusion imaging at the discretion of the family physician or primary cardiologist.

These follow up LVEF measurements will be entered into the APPROACH database in order to allow us to evaluate the clinical significance of changes in EF after MI and prognostic significance of initial versus follow-up EF values.

Data Analysis

AMIQA Phase I: Quality Assurance

Data collected will be entered into a database and summary statistics will be created (e.g. proportion of follow up LVEF assessments completed post-MI (Aim 5.1), choice of modality for follow up LVEF assessment, etc.) Data collected from the surveys will be entered into a database and analyzed in SAS or Stata. Summary statistics will be created from the data collected in the surveys.

Acute Myocardial Infarction Quality Assurance (AMIQA) Project Research Protocol - Updated Feb 29, 2012

AMIQA Phase II: Prognostic Factor Study

As part of AMIQA Phase II, LVEF assessments will be entered into the APPROACH database. The study will compare initial LVEF measurements post-MI to follow-up LVEF measurements, and assess for improvement, stability and deterioration of LVEF and the factors associated with these changes in LVEF.

This project has received ethics approval by the Conjoint Health Research and Ethics Board of the University of Calgary. Patients will be identified using the APPROACH database have provided written, informed consent as part of their participation in APPROACH. Only the research team will know the names and contact information of the patients included in the study, and this information will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* confirmed MI

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients surviving an acute MI.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 years

SECONDARY OUTCOMES:
Ejection Fraction | 12 months
Heart Failure Hospitalization | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Derek V Exner, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada